CLINICAL TRIAL: NCT05687266
Title: A Phase III, Randomised, Open-label, Multicentre, Global Study of Datopotamab Deruxtecan (Dato-DXd) in Combination With Durvalumab and Carboplatin Versus Pembrolizumab in Combination With Platinum-based Chemotherapy for the First-line Treatment of Patients With Locally Advanced or Metastatic NSCLC Without Actionable Genomic Alterations (D926NC00001; AVANZAR)
Brief Title: Phase III, Open-label, First-line Study of Dato-DXd in Combination With Durvalumab and Carboplatin for Advanced NSCLC Without Actionable Genomic Alterations
Acronym: AVANZAR
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D926NC00001; 2021-004606-21 (EudraCT Number)
Record Dates: First submitted 2022-12-28; First posted 2023-01-18 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: NSCLC
Keywords: Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC); Datopotamab deruxtecan (Dato-DXd, Datroway); Durvalumab (Imfinzi); Carboplatin; Chemotherapy; Antibody-Drug Conjugate (ADC); Trophoblast cell surface protein 2 (TROP2)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; Carboplatin; pembrolizumab; Cisplatin; Pemetrexed; Paclitaxel

STUDY DESIGN:
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dato-DXd + Durvalumab + Carboplatin (Experimental): Participants will be randomized to receive 6.0mg/kg Dato-DXd plus 1120 mg durvalumab plus carboplatin area under the curve [AUC] 5 mg/mL/minute.
  Interventions: Drug: Datopotamab deruxtecan; Drug: Durvalumab; Drug: Carboplatin
- Histologic-specific therapy (Active Comparator): Non-squamous NSCLC participants will be randomized to receive 200 mg pembrolizumab plus 500 mg/m2 pemetrexed plus either AUC 5 mg/mL/minute carboplatin or 75 mg/m2 cisplatin.
  Squamous NSCLC participants will be randomized to receive 200 mg of pembrolizumab plus 200 mg/m2 paclitaxel plus AUC 5 or 6 mg/mL/minute carboplatin.
  Interventions: Drug: Carboplatin; Drug: Pembrolizumab; Drug: Cisplatin; Drug: Pemetrexed; Drug: Paclitaxel

INTERVENTIONS:
Drug: Datopotamab deruxtecan — Intravenous (IV) infusion every 3 weeks (Q3W) on Day 1 of each 21-day cycle.
  Other Names: Dato-DXd, Datroway
  Arms: Dato-DXd + Durvalumab + Carboplatin
Drug: Durvalumab — Intravenous (IV) infusion every 3 weeks (Q3W) on Day 1 of each 21-day cycle.
  Other Names: MEDI4736, Imfinzi
  Arms: Dato-DXd + Durvalumab + Carboplatin
Drug: Carboplatin — Intravenous (IV) infusion every 3 weeks on Day 1 of each 21-day cycle for up to 4 cycles.
Drug: Pembrolizumab — Intravenous (IV) infusion every 3 weeks (Q3W) on Day 1 of each 21-day cycle for a maximum of 35 cycles or 2 years (whichever occurs first).
  Arms: Histologic-specific therapy
Drug: Cisplatin — Intravenous (IV) infusion every 3 weeks on Day 1 of each 21-day cycle for up to 4 cycles.
  Arms: Histologic-specific therapy
Drug: Pemetrexed — Intravenous (IV) infusion every 3 weeks on Day 1 of each 21-day cycle.
  Arms: Histologic-specific therapy
Drug: Paclitaxel — Intravenous (IV) infusion every 3 weeks on Day 1 of each 21-day cycle for up to 4 cycles.
  Arms: Histologic-specific therapy

SUMMARY:
This is a Phase III, randomized, open-label, multicenter, global study to compare the efficacy and safety of Datopotamab Deruxtecan (Dato-DXd) in combination with durvalumab and carboplatin compared with pembrolizumab in combination with histology-specific platinum-based chemotherapy as first-line treatment of adults with stage IIIB, IIIC, or IV NSCLC without actionable genomic alterations (including sensitizing EGFR mutations, and ALK and ROS1 rearrangements).

DETAILED DESCRIPTION:
Participants with locally advanced or metastatic NSCLC without actionable tumor tissue genomic alterations and confirmed to meet all eligibility criteria will be randomized in a 1:1 ratio to Dato-DXd in combination with durvalumab and carboplatin versus pembrolizumab in combination with histology-specific platinum-based chemotherapy as first-line treatment.

The primary objectives of the study are to demonstrate superiority of Dato-DXd in combination with durvalumab and carboplatin relative to pembrolizumab in combination with platinum-based chemotherapy by assessment of the following:

1. PFS by BICR in first-line treatment of participants with non-squamous TROP2 biomarker positive locally-advanced or metastatic NSCLC
2. OS in first-line treatment of participants with non-squamous TROP2 biomarker positive locally-advanced or metastatic NSCLC
3. PFS by BICR in first-line treatment of participants with non-squamous locally-advanced or metastatic NSCLC
4. OS in first-line treatment of participants with non-squamous locally-advanced or metastatic NSCLC

ELIGIBILITY:
Inclusion:

* Participants ≥ 18 years at screening
* Histologically or cytologically documented NSCLC that at the time of randomisation is Stage IIIB or IIIC disease not amenable to surgical resection or definitive chemoradiation or Stage IV metastatic disease
* Lacks sensitising EGFR tumour tissue mutation and ALK and ROS1 rearrangements and has no documented tumour genomic alterations in NTRK, BRAF, RET, MET or other actionable driver oncogenes with approved and available therapies (actionable genomic alterations).

Testing is not required for tumors with squamous histology, with exceptions.

* ECOG PS of 0 or 1
* Archival tumour tissue
* Has adequate bone marrow reserve and organ function within 7 days before randomization

Exclusion:

* Mixed small-cell lung cancer and NSCLC histology; sarcomatoid variant of NSCLC
* History of another primary malignancy with exceptions
* Persistent toxicities caused by previous anti-cancer therapy not yet improved to Grade ≤ 1 or baseline, with exceptions.
* Spinal cord compression or clinically or radiologically active brain metastases
* History of leptomeningeal carcinomatosis.
* Known active or uncontrolled hepatitis B or C virus infection.
* Uncontrolled or suspected infection requiring IV antibiotics, antivirals, or antifungals.
* Clinically significant corneal disease
* History of non-infectious ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or has suspected ILD/pneumonitis that cannot be ruled out by imaging at screening.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1350 (Actual)
Dates: Start 2022-12-29 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) by blinded independent central review (BICR) in the non-squamous TROP2 biomarker positive population | Approximately 3 years
  PFS is deﬁned as time from randomisation until progression per Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1) as assessed by BICR, or death due to any cause.
Overall Survival (OS) in the non-squamous TROP2 biomarker positive population | Approximately 5 years
  OS is defined as the time from randomisation until the date of death due to any cause.
PFS by BICR in the non-squamous population | Approximately 3 years
  PFS is deﬁned as time from randomisation until progression per RECIST 1.1 as assessed by BICR, or death due to any cause.
OS in the non-squamous population | Approximately 5 years
  OS is deﬁned as the time from randomisation until the date of death due to any cause.

SECONDARY OUTCOMES:
PFS by BICR in ITT and TROP2 biomarker-defined populations | Approximately 3 years
  PFS is defined as time from randomisation until progression per RECIST 1.1 as assessed by BICR, or death due to any cause.
OS in ITT and TROP2 biomarker-defined populations | Approximately 5 years
  OS is defined as the time from randomisation until the date of death due to any cause.
Objective Response Rate (ORR) in ITT, non-squamous and TROP2 biomarker-defined populations | Approximately 5 years
  ORR is deﬁned as the proportion of participants who have a conﬁrmed Complete Response (CR) or conﬁrmed Partial Response (PR), as determined by BICR per RECIST 1.1.
Duration of Response (DoR) in ITT, non-squamous and TROP2 biomarker-defined populations | Approximately 5 years
  DoR is deﬁned as the time from the date of ﬁrst documented conﬁrmed response until date of documented progression per RECIST 1.1, as assessed by BICR and investigator clinical assessment or death due to any cause.
PFS by investigator in ITT, non-squamous and TROP2 biomarker-defined populations | Approximately 3 years
  PFS is deﬁned as time from randomisation until progression per RECIST 1.1 as assessed by investigator clinical assessment, or death due to any cause.
Pharmacokinetics of Dato-DXd when combined with durvalumab and carboplatin. | Approximately 5 years
  Concentration of Dato-DXd, total anti-TROP2 antibody, and DXd (payload deruxtecan) in plasma and pharmacokinetic (PK) parameters (such as peak and trough concentrations, as data allow; sparse sampling).
Anti-Drug Antibody (ADA) for Dato-DXd | Approximately 5 years
  The immunogenicity of Dato-DXd when combined with durvalumab and carboplatin.
Time to Second Progression or Death (PFS2) in ITT, non-squamous and TROP2 biomarker-defined populations | Approximately 5 years
  PFS2 is defined as the time from randomisation to the earliest of the progression events (following the initial progression), subsequent to first subsequent therapy, or death.
Clinical Outcome Assessments in ITT, non-squamous and TROP2 biomarker-defined populations | Approximately 5 years
  Clinical Outcome Assessments, such as TTD in pulmonary symptoms (dyspnoea, cough and chest pain) as measured by the NSCLC-SAQ, and TTD in physical functioning as measured by PROMIS Physical Function short form 8c

OTHER OUTCOMES:
Safety of Dato-DXd in combination with durvalumab and carboplatin | Approximately 5 years
  Safety and tolerability will be evaluated in terms of AEs (graded by CTCAE Version 5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Charu Aggarwal, Study Chair — Perelman Center for Advanced Medicine
Locations (214):
- United States (48):
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Hot Springs, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Springdale, Arkansas
  - Research Site, Fountain Valley, California
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, Boulder, Colorado
  - Research Site, Fort Myers, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Hinsdale, Illinois
  - Research Site, Fort Wayne, Indiana
  - Research Site, Bettendorf, Iowa
  - Research Site, Iowa City, Iowa
  - Research Site, Waukee, Iowa
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Covington, Louisiana
  - Research Site, Duluth, Minnesota
  - Research Site, Rochester, Minnesota
  - Research Site, Hannibal, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Clifton Park, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Maumee, Ohio
  - Research Site, Tulsa, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Salem, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, York, Pennsylvania
  - Research Site, Watertown, South Dakota
  - Research Site, Memphis, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Irving, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, Henrico, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Renton, Washington
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Appleton, Wisconsin
  - Research Site, La Crosse, Wisconsin
- Austria (3):
  - Research Site, Graz
  - Research Site, Rankweil
  - Research Site, Vienna
- Brazil (8):
  - Research Site, Blumenau
  - Research Site, Florianópolis
  - Research Site, Fortaleza
  - Research Site, Londrina
  - Research Site, Porto Alegre
  - Research Site, São Paulo
  - Research Site, Taubaté
  - Research Site, Vitória
- Bulgaria (2):
  - Research Site, Sofia
  - Research Site, Varna
- Canada (8):
  - Research Site, Saint John, New Brunswick
  - Research Site, Brampton, Ontario
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Kitchener, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Saint-Jérôme, Quebec
  - Research Site, Saskatoon, Saskatchewan
- China (22):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Kunming
  - Research Site, Lanzhou
  - Research Site, Liuchow
  - Research Site, Shandong
  - Research Site, Shanghai
  - Research Site, Shantou
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xiamen
  - Research Site, Yangzhou
  - Research Site, Zhengzhou
- France (12):
  - Research Site, Brest
  - Research Site, Créteil
  - Research Site, Gleizé
  - Research Site, Montpellier
  - Research Site, Nîmes
  - Research Site, Paris
  - Research Site, Rouen
  - Research Site, Saint-Quentin
  - Research Site, Strasbourg
  - Research Site, Toulon
  - Research Site, Toulouse
  - Research Site, Tours
- Germany (13):
  - Research Site, Bad Berka
  - Research Site, Berlin
  - Research Site, Frankfurt A. Main
  - Research Site, Gauting
  - Research Site, Gütersloh
  - Research Site, Hamburg
  - Research Site, Kassel
  - Research Site, Kiel
  - Research Site, Koblenz
  - Research Site, Minden
  - Research Site, Rosenheim
  - Research Site, Velbert
  - Research Site, Würzburg
- Greece (3):
  - Research Site, Athens
  - Research Site, Piraeus
  - Research Site, Thessaloniki
- Hungary (7):
  - Research Site, Budapest
  - Research Site, Gyöngyös - Mátraháza
  - Research Site, Kaposvár
  - Research Site, Pécs
  - Research Site, Szekszárd
  - Research Site, Szolnok
  - Research Site, Törökbálint
- India (6):
  - Research Site, Calicut
  - Research Site, Delhi
  - Research Site, Jaipur
  - Research Site, Kolkata
  - Research Site, Madurai
  - Research Site, Puducherry
- Italy (9):
  - Research Site, Florence
  - Research Site, Lecco
  - Research Site, Messina
  - Research Site, Napoli
  - Research Site, Orbassano
  - Research Site, Padua
  - Research Site, Parma
  - Research Site, Peschiera del Garda
  - Research Site, Rozzano
- Japan (15):
  - Research Site, Bunkyō City
  - Research Site, Chūōku
  - Research Site, Hamamatsu
  - Research Site, Hidaka-shi
  - Research Site, Hirosaki-shi
  - Research Site, Hiroshima
  - Research Site, Kumamoto
  - Research Site, Nagoya
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Sapporo
  - Research Site, Sunto-gun
  - Research Site, Wakayama
  - Research Site, Yokohama
- Mexico (4):
  - Research Site, Del. Cuauhtemoc
  - Research Site, Mexico City
  - Research Site, México
  - Research Site, San Luis Potosí City
- Peru (3):
  - Research Site, Arequipa
  - Research Site, Concepción
  - Research Site, Lima
- Poland (11):
  - Research Site, Bydgoszcz
  - Research Site, Bystra
  - Research Site, Grudziądz
  - Research Site, Kielce
  - Research Site, Koszalin
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Przemyśl
  - Research Site, Racibórz
  - Research Site, Radom
  - Research Site, Siedlce
- South Korea (5):
  - Research Site, Busan
  - Research Site, Cheongju-si
  - Research Site, Jinju
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (7):
  - Research Site, Las Palmas de Gran Canaria
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Santander
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Zaragoza
- Sweden (5):
  - Research Site, Gävle
  - Research Site, Linköping
  - Research Site, Lund
  - Research Site, Stockholm
  - Research Site, Uppsala
- Taiwan (6):
  - Research Site, Hsinchu
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Turkey (Türkiye) (5):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Edirne
  - Research Site, Istanbul
  - Research Site, Izmir
- United Kingdom (10):
  - Research Site, Aberdeen
  - Research Site, Cambridge
  - Research Site, Cardiff
  - Research Site, Cheltenham
  - Research Site, Edinburgh
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Middlesbrough
  - Research Site, Newcastle upon Tyne
  - Research Site, Taunton
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/